CLINICAL TRIAL: NCT05686980
Title: An Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ABBV-552 in Healthy Adult Japanese and Han Chinese Subjects
Brief Title: A Study to Assess the Adverse Events and How Oral ABBV-552 Capsules Moves Through the Body of Healthy Adult Japanese and Han Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23-512
Record Dates: First submitted 2023-01-13; First posted 2023-01-17 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
Keywords: ABBV-552; Alzheimer's disease (AD)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Healthy Japanese Participants (Experimental): Participants will receive ABBV-552 once a week for 21 Days.
  Interventions: Drug: ABBV-552
- Arm 2: Healthy Han Chinese Participants (Experimental): Participants will receive ABBV-552 once a week for 7 Days.
  Interventions: Drug: ABBV-552

INTERVENTIONS:
Drug: ABBV-552 — Oral Capsule

SUMMARY:
This study will assess how safe ABBV-552 is and how ABBV-552 moves through the body of adult healthy Japanese and Han Chinese participants. Adverse Events will be assessed.

ABBV-552 is an investigational drug being developed for potential treatment of Alzheimer's disease (AD). Approximately 18 adult healthy Japanese and Han Chinese volunteers will be enrolled in 2 sites in the United States.

Japanese participants assigned to Arm 1 will receive ascending doses of ABBV-552 oral capsules once every week for 3 weeks. Han Chinese participants assigned to Arm 2 will receive oral ABBV-552 capsules on Day 1. All participants will be followed for 30 days after their last dose.

Participants will be confined for 22 days or 8 days depending on the Arm they are assigned to. Adverse Events and blood tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

- Japanese participants must be first- or second-generation Japanese of full Japanese parentage. First-generation participants will have been born in Japan to two parents and four grandparents also born in Japan of full Japanese descent. Second-generation participants born outside of Japan must have two parents and four grandparents born in Japan of full Japanese descent. All participants must maintain a typical Japanese lifestyle, including consuming a typical Japanese diet.

OR

* Han Chinese participants must be first-generation Han Chinese of full Chinese parentage residing outside of China for less than 5 years. Participants must maintain a typical Chinese lifestyle, including consuming a typical Chinese diet.

Exclusion Criteria:

- Has no other clinically significant and/or unstable medical conditions or any other reason that the investigator determines would interfere with the participant's participation in this study or would make the participant an unsuitable candidate to receive ABBV-552.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AE) | Up to approximately 45 days
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Plasma Concentration (Cmax) of ABBV-552 | Up to approximately 21 days
  Maximum observed plasma concentration (Cmax) of ABBV-552.
Time to Cmax (Tmax) of ABBV-552 | Up to approximately 21 days
  The time to Cmax (Tmax) of ABBV-552.
Terminal Phase Elimination Rate Constant (λz) of ABBV-552 | Up to approximately 21 days
  Terminal phase elimination rate constant (λz) of ABBV-552.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-552 | Up to approximately 21 days
  Terminal phase elimination half-life (t1/2) of ABBV-552.
Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to the Last Measurable Concentration (AUCt) of ABBV-552 | Up to approximately 21 days
  AUCt of ABBV-552.
AUC From Time Zero to Infinite Time (AUCinf) of ABBV-552 | Up to approximately 21 days
  AUCinf of ABBV-552.
Apparent Oral Clearance (CL/F) of ABBV-552 | Up to approximately 21 days
  Apparent oral clearance (CL/F) of ABBV-552.
Apparent Volume of Distribution (Vz/F) of ABBV-552 | Up to approximately 21 days
  Apparent volume of distribution (Vz/F) of ABBV-552.
Dose-Normalized Cmax of ABBV-552 (Arm 1) | Up to approximately 21 days
  Dose-normalized Cmax of ABBV-552.
AUC of ABBV-552 (Arm 1) | Up to approximately 21 days
  AUC of ABBV-552.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Anaheim Clinical Trials LLC /ID# 252203, Anaheim, California
  - PPD Clinical Research Unit -Las Vegas /ID# 252241, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-512